CLINICAL TRIAL: NCT06904144
Title: Health Coaching for Patients With Cardiovascular Disease: A Mixed-Methods Evaluation of the Impact on Patient Outcomes and Provider Satisfaction and Acceptability
Brief Title: Health Coaching for Patients With Cardiovascular Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Beth Steinberg, Associate Director of Research, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024H0179
Record Dates: First submitted 2025-03-03; First posted 2025-04-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Congestive Heart Failure Treated; Myocardial Infarction (MI); Coronary Artery Disease; Congestive Heart Failure Chronic
Keywords: health coaching; coronary artery disease; congestive heart failure; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching Intervention Group (Experimental): Participants will receive 12 health coaching sessions post-discharge over a 16 week period
  Interventions: Behavioral: Health Coaching
- Standard Care Group (No Intervention): Participants will receive usual post-discharge care over the 16 week period

INTERVENTIONS:
Behavioral: Health Coaching — 12 virtual health coaching sessions will be provided over a 16 week period by a certified health coach.
  Arms: Health Coaching Intervention Group

SUMMARY:
For patients discharged with a diagnosis of cardiovascular disease coronary artery disease resulting in myocardial infarction and/or congestive heart failure, this study will evaluate if the addition of 12 virtual health coaching sessions over the course of 16 weeks will improve physiological, psychological, and social health outcomes, prove acceptable and satisfactory for these patients with CVD, decrease CVD-related questions and concerns sent to the provider via MyChart, and reduce hospital readmission rates over a 90-day period as compared to patients discharged with the same diagnosis who receive standard post-discharge care. The study will also evaluate the perceptions of physician and advanced practice providers related to the health coach as part of the interprofessional team and the amount of time spent addressing CVD-related patient questions and concerns via MyChart messages.

DETAILED DESCRIPTION:
The purpose of this mixed methods study is to evaluate the impact of 12 virtual health coaching sessions, provided post-discharge, over the course of 16 weeks on: 1) patient physiological measure of weight; 2) patient-reported perceived stress, anxiety, depression, and medication adherence, and physical, emotional, and social lifestyle behaviors; and 3) MyChart messaging to their providers related to concerns and/or questions about their cardiovascular diagnosis. The study will also assess: 4) patient acceptability and satisfaction with the health coaching intervention; 5) acceptability and satisfaction value and/or importance of the health coach intervention and feasibility of integrating the health coach into the inter-professional care team from the provider perspective; impact of the health coaching intervention on provider time spent on addressing MyChart messages; and 6) 30-, 60-, and 90-day hospital readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* diagnosis of coronary artery disease resulting in myocardial infarction and/or congestive heart failure
* physical condition effectively managed by routine healthcare and not requiring urgent medical attention
* ability to communicate in English
* access to a working phone or computer and ability to communicate via phone or computer.

Exclusion Criteria:

* Patients who have had chest coronary artery bypass surgery
* Documented cognitive and/or major psychiatric disorders, including dementia, Alzheimer's, depression or anxiety uncontrolled by anxiolytic, anti-psychotic, and/or anti-depressants and/or PHQ-9 score 15-27 and GAD-7 score >15
* current alcohol or drug dependency
* resident of extended care/skilled facility
* prisoners or ward of state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | Baseline (day of hospital discharge) and at provider appointment in the ambulatory setting, 16 weeks post-hospital discharge
  Patient body weight in kilograms will be obtained by clinical staff on hospital approved and calibrated electronic standing scales. The patient's body weight will be collected from the patient's electronic medical record.
Hospital readmissions | Hospital readmissions during the 30-, 60-, and 90-days post-hospital discharge for cardiovascular disease, documented in the electronic medical record
  Hospital readmissions for an inpatient stay, documented in the electronic medical record, after the hospital post-discharge for cardiovascular disease
MyChart messages | Over the course of 16 weeks, from hospital discharge to 16 weeks post-hospital discharge
  MyChart messages are questions or requests directed to the patient's provider that are related to the patient's cardiovascular disease diagnosis and hospitalization. These MyChart messages are entered into the electronic medical record by the patient and are directed to their provider, requiring an electronic or telephone response to the patient with a documented note entered by the provider relative to the follow-up provided to the patient. This outcome measure will be the number of MyChart messages entered by the patient and responded to by the provider.
Perceived Stress | Baseline (hospital discharge), 8 weeks post-hospital discharge, and 16 weeks post-hospital discharge
  Perceived Stress Scale-10 (PSS-10). A 10-item self-report measure of perceived stress. It is a measure of the degree to which situations in one's life are appraised as stressful over the past month. The 4-point Likert Scale includes responses of 0 (never), 1 (almost never), 2 (sometimes), 3 (fairly often), and 4 (very often). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Medication Adherence | Baseline, and at 8 weeks post-hospital discharge and at 16 weeks post-hospital discharge
  The Hill-Bone Medication Adherence Scale (MB-MAS) is a 9-item self-assessment of medication adherence relative to a variety of chronic diseases and conditions. Likert Scale responses to each of the nine statements include 1 (all of the time), 2 (most of the time), 3 (some of the time), and 4 (none of the time). Total scores range from 4 to 36 with higher scores indicating higher medication adherence.
Lifestyle Medicine Behavior Assessment | Completed at baseline, at 8 weeks post-hospital discharge and at 16 weeks post-hospital discharge
  The Lifestyle Medicine Short Form is a 14-item self-assessment scale evaluating physical, emotional, social lifestyle behaviors. The assessment questions comprise core metrics that capture readiness to change, as well as health behaviors that are aligned with the six pillars of lifestyle medicine--physical activity, nutrition, sleep health, stress reduction, social connections, and risky substances. Questions have multiple responses based on information relating to the six pillars of lifestyle medicine. The first two questions related to Readiness to Change use a Likert Scale ranging from 0 (Not Ready) to 10 (Very Ready). Questions related to Motivation and Diet request that the participant denote different aspects of their diet. Physical exercise questions request specific days/times in minutes completed. Questions related to sleep request average hours of sleep per 24 hour period. Mood, connectedness with others, and substance use request types/amounts per week.
Acceptability of Intervention Measure | Completed after the 16 week health coaching intervention for participants in the intervention group.
  The Acceptability of Intervention Measure (AIM) is a 4-item self-report assessment to evaluate the acceptability of the health coaching intervention. Each statement is scored with a 5-point Likert Scale that includes 1 (completely disagree), 2 (disagree), 3 (neither agree nor disagree), 4 (agree), and 5 (completely agree). Total scores ranges from 4-20 with higher total scores indicating higher acceptability.

SECONDARY OUTCOMES:
Patient Qualitative Comments | Immediately after completion of the 16 week health coaching intervention; i.e. 16 weeks post-hospital discharge
  Patient perceptions of the health coaching intervention will be solicited with the following question prompts: 1) Can you provide feedback about your health coaching experience?; 2) Did working with the health coach help you meet your health goals?; 3) Would you recommend working with a health coach to others?
Provider Qualitative Comments | Will be completed within one month of their patient completing the health coach intervention.
  Provider perceptions of the value of the health coach as part of the interprofessional team and the feasibility of integrating the health coach into the patient's care will be solicited via question prompts that will include: 1) Can you discuss your perceptions about the value of the health coach as a member of the patient's care team; 2) Were you able to review the health coaches notes in the patient's medical record? (if yes) Were the notes helpful to you during the patient's follow-up appointment(s), i.e. in addressing the patient's condition, their post-discharge recovery, adherence to medical instructions, progress or lack of progress?; 3) Can you provide your perceptions of the feasibility of integrating the health coach as part of the patient's care team?
Patient Health Questionnaire (PHQ-9) | Baseline, 4-, 8-, and 16 weeks post-discharge for all participants
  A 9-item depression module the Patient Health Questionnaire that scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day); scores range from 9-27.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 4-, 8-, and 16 weeks post-discharge for all participants
  A 7-item screening tool assessing anxiety over the past 2 weeks. Questions are scored from "0" (not at all) to "3" (nearly every day). Scores range from 0-21.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Steinberg, PhD, RN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that will be shared will include de-identified descriptive data for both the intervention and control groups, including gender, race, educational level and mean age. Additionally, cardiovascular disease diagnoses, hospital readmissions at 30-, 60-, and 90- days post-hospital discharge, and number of MyChart messages sent by the patient to their provider. Acceptability of the intervention descriptive data for the intervention group will also be included. Differences in mean scores between the intervention and control groups for weight (significance and effect sizes), perceived stress and medication adherence will be shared. De-identified, curated qualitative data that will be shared includes interview transcripts from both patients and providers, as well as the qualitative codebooks and thematic analysis.
Supporting Information: ICF, CSR, Analytic Code
Time Frame: 12-30-2026 to indefinitely
Access Criteria: De-identified and curated demographic, statistical data, study overview, study consent will be accessible to academic researchers and educators through a data accessibility link once the Qualitative Data Repository submission is finalized.